CLINICAL TRIAL: NCT05661682
Title: A Randomized, Single-blind, Trial of Tralement Versus a Fixed-dose Trace Element Combination Product of Zinc, Copper, and Selenious Acid to Evaluate Manganese Safety in Adult Patients Requiring Long-term Parenteral Nutrition
Brief Title: Tralement Versus a Fixed-dose Trace Element Combination Product to Evaluate Manganese Safety
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: American Regent, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TE20001
Record Dates: First submitted 2022-12-13; First posted 2022-12-22 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Manganese Safety in Adults
MeSH Terms: interventions — manganese sulfate; Zinc Sulfate; Copper Sulfate; Selenious Acid; Copper; Zinc

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tralement (Active Comparator): This study will enroll new prescribed home parenteral nutrition users, i.e. a patient enrolled in the study within six weeks of initiating first-time use of parenteral nutrition formulation requiring trace element additives. Note: a portion of patients who meet inclusion criteria may have received parenteral nutrition in an inpatient setting before discharge home.
  Interventions: Drug: Tralement
- a fixed-dose trace element combination product of zinc sulfate, copper sulfate, and selenious acid (Active Comparator): This study will enroll new prescribed home parenteral nutrition users, i.e. a patient enrolled in the study within six weeks of initiating first-time use of parenteral nutrition formulation requiring trace element additives. Note: a portion of patients who meet inclusion criteria may have received parenteral nutrition in an inpatient setting before discharge home.
  Interventions: Drug: Fixed-dose trace element combination product of zinc, copper, and selenious acid

INTERVENTIONS:
Drug: Tralement — Tralement with Manganese Sulfate
  Other Names: manganese sulfate, zinc sulfate, copper sulfate, and selenious acid
  Arms: Tralement
Drug: Fixed-dose trace element combination product of zinc, copper, and selenious acid — Tralement without Manganese Sulfate
  Other Names: zinc, copper, and selenious acid
  Arms: a fixed-dose trace element combination product of zinc sulfate, copper sulfate, and selenious acid

SUMMARY:
Tralement versus a fixed-dose trace element combination product of zinc, copper, and selenious acid to evaluate product safety in adult patients requiring long-term parenteral nutrition.

DETAILED DESCRIPTION:
A Phase IV, multi-center, randomized single-blind trial to evaluate the safety profile of Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid in adult patients who are expected to require at least six-months of home parenteral nutrition.

This study will enroll new prescribed home parenteral nutrition users, i.e. a patient enrolled in the study within six weeks of initiating first-time use of parenteral nutrition requiring trace element additives. Note: a portion of patients who meet inclusion criteria may have received parenteral nutrition in an inpatient setting before discharge home.

Eligible participants who satisfy the inclusion requirements and no exclusion criteria will be consented to participate in this study and enter the screening study phase.

The screening evaluation will be conducted within 5 days of the dose administration of study drug. Study participants meeting entry criteria of normal brain MRI and laboratory manganese concentrations (whole blood/plasma/serum/RBC) will begin study drug on Day 1.

Participants will undergo 2 additional post-baseline brain MRI scans at Months 3 and 6 and have 5 separate neuropsychological tests at Day 1, Month 3, and Month 6. Additional clinical monitoring including safety and laboratory assessments will occur during the 6-month opt-in extension study.

All patients in each assigned trace element parenteral nutrition group will have parenteral nutrition formulations evaluated for manganese content at Day 1, Month 1, Month 3, and Month 6.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 to ≤80 years of age) participants able to provide informed consent.
* Male and female participants who are new users to home parenteral nutrition as a source of trace elements when oral or enteral nutrition is not possible, insufficient, or, contraindicated.
* Anticipated duration of home parenteral nutrition use is 6 months or greater.
* A normal baseline brain MRI scan.
* A normal blood manganese concentration.
* Ability to undergo additional 2 brain MRI scans over the six-month study period (Sedation, if appropriate, to be determined by the Principal Investigator's study site, institutional review board recommendations).
* Definitive contraception for females of reproductive age.

Exclusion Criteria:

* Prior parenteral nutrition therapy.
* Hypersensitivity or allergy to zinc or copper.
* History of occupational exposure to manganese and documented by laboratory test results.
* Baseline ferritin ≥300 ng/mL or below 100 ng/mL.
* Baseline transferrin saturation (TSAT) ≥45 % or below 20%.
* Prior or current cholestatic liver disease defined as a clinical condition associated with decrease in bile flow due to impaired secretion by hepatocytes or to obstruction of bile flow through intra-or extrahepatic bile ducts.
* Liver function studies with transaminases greater than two-fold normal or total bilirubin >2 mg/dL.
* Brain MRI exclusion criteria: MRI-unsafe metal implants, claustrophobia.
* Known excess environmental exposure to manganese.
* Less than 1-year expected survival, as anticipated by their primary provider.
* Current participation in another clinical trial.
* Females in pregnant state.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2026-12-04 (Estimated)

PRIMARY OUTCOMES:
To assess brain deposition of manganese in Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid. | 6 Months
  Change from baseline in basal ganglia index (BG-index) as determined by T1-weighted brain MRI images.

SECONDARY OUTCOMES:
To assess the efficacy & safety of Tralement versus a fixed-dose trace element product of zinc, copper, and selenious acid. | 6 Months
  Change from baseline in blood (plasma/serum/RBC) manganese levels assessed

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Khechen, MD, Study Director — Sr. Medical Director